CLINICAL TRIAL: NCT06151834
Title: Prospective Study of Arthrodesis of Finger Distal Interphalangeal Joints Using the Kerifuse Device KF 23)
Brief Title: Prospective Study of Arthrodesis of Finger Distal Interphalangeal Joints Using the Kerifuse Device
Acronym: KF23
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Clinique Saint François, Nice, France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-A02072-43
Record Dates: First submitted 2023-11-14; First posted 2023-11-30 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Osteoarthritis Finger; Osteoarthritis Thumb

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients (Experimental): Patients older than 18 years-old, with a surgical indication of interphalangeal arthrodesis of finger
  Interventions: Procedure: KeriFuse implant implantation

INTERVENTIONS:
Procedure: KeriFuse implant implantation — The surgery is an arthrodesis of finger or thumb (for patients with finger osteoarthritis) and involves implanting the KeriFuse implant.

SUMMARY:
Arthrodesis of a distal interphalangeal joint of the finger (DIP) is mainly performed for a degenerated and painful joint. Various stabilization methods have been used to provide compression at the arthrodesis site such as pins, steel wires, compression screws, headless compression screws, bioresorbable implants and intramedullary staples.

Although with complications such as implant fractures or dorsal cortical erosion, intramedullary arthrodesis staples provide reliable pain relief and a consistent fusion rate while inevitably scarring the finger pulp or nail dystrophy.

The aim of this study is to evaluate the bone fusion time during an arthrodesis performed with the Kerifuse shape memory implant.

DETAILED DESCRIPTION:
Arthrodesis of a distal interphalangeal joint of the finger (DIP) is mainly performed for a degenerated and painful joint. Various stabilization methods have been used to provide compression at the arthrodesis site such as pins, steel wires, compression screws, headless compression screws, bioresorbable implants and intramedullary staples.

Although with complications such as implant fractures or dorsal cortical erosion, intramedullary arthrodesis staples provide reliable pain relief and a consistent fusion rate while inevitably scarring the finger pulp or nail dystrophy.

The aim of this study is to evaluate the bone fusion time during an arthrodesis performed with the Kerifuse shape memory implant.

Main objective is to evaluate the bone fusion time in arthrodesis performed with the Kerifuse shape memory implant.

Secondary objectives are :

* to evaluate the fusion rate and its associated healing time
* to evaluate patient satisfaction, including aesthetic aspect
* to assess overall hand function
* to evaluate the radiological evolution of the KeriFuse® implant and its implantation site
* To evaluate the radiological evolution of the arthrodesis angle between the post-operative situation and the final fusion position

ELIGIBILITY:
Inclusion Criteria:

* Eligible patients with osteoarthritis of finger for an interphalangeal arthrodesis with KeriFuse implant

Exclusion Criteria:

* Pregnant or breastfeeding patient
* Patient with an intellectual disability and who therefore cannot follow the surgeon's instructions
* Patients with contraindications to surgery
* Patients with acute or chronic, local or systemic infections
* Patients with sensitivities or allergies to device components (Nickel, Titanium)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Fusion time of bone in distal interphalangeal arthrodesis of the fingers | day 5 - week 4 - week 6 - week 8 - week 10 - week 12 - year 2 after surgery
  Fusion time of bone (in weeks) will be measure by X-ray,

SECONDARY OUTCOMES:
Mid-term efficacy of arthrodesis in pain decrease | day 5 - week 4 - week 6 - week 8 - week 10 - week 12 - year 2 after surgery
  Evaluation of pain with analogic visual scale
Evaluation of arthrosis degree | day 5 - week 4 - week 6 - week 8 - week 10 - week 12 - year 2 after surgery
  Evaluation fo arthrosis degree according to Kellgren-Lawrence scale
Patient satisfaction | D5 - W4 - W6 - W8 - W10 - W12 - Y2 after surgery
  Evaluation of patient satisfaction according to Likert scale
Evaluation of global hand function | day 5 - week 4 - week 6 - week 8 - week 10 - week 12 - year 2 after surgery
  Evaluation by the patient using functional score Quick DASH

CONTACTS AND LOCATIONS:
Locations (1):
- Clinique Saint François, Nice, France

IPD SHARING:
Plan to Share IPD: No